CLINICAL TRIAL: NCT03017443
Title: Effects of a Commercially-Available Structured Weight Loss Program Provided in Three Different Formats on Anthropometric Measures in Healthy Overweight and Obese Adults
Brief Title: Study to Evaluate Effects of a Weight Loss Program in Different Formats on Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nutrisystem, Inc. (Industry)
Collaborators: Biofortis Clinical Research, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIO-1507
Record Dates: First submitted 2017-01-06; First posted 2017-01-11 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 2017-01

CONDITIONS: Overweight and Obesity; Weight Loss
Keywords: Weight Loss; Obesity; Overweight
MeSH Terms: conditions — Overweight; Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Nutrisystem My Way (Experimental): All subjects received Nutrisystem pre-packaged, portion-controlled foods and followed the Nutrisystem My Way plan.
  Interventions: Behavioral: Nutrisystem My Way
- Nutrisystem Turbo 10 (Experimental): All subjects received Nutrisystem pre-packaged, portion-controlled foods and followed the Nutrisystem Turbo 10 plan.
  Interventions: Behavioral: Nutrisystem Turbo 10
- Nutrisystem DASH (Experimental): All subjects received Nutrisystem pre-packaged, portion-controlled foods and followed the Nutrisystem DASH plan.
  Interventions: Behavioral: Nutrisystem DASH
- Dieting on Your Own (DIY) - DASH (Active Comparator): All subjects provided publically available information on the DASH diet and instructed to follow a reduced calorie DASH diet meal plan on their own.
  Interventions: Behavioral: Dieting on Your Own (DIY) - DASH

INTERVENTIONS:
Behavioral: Nutrisystem Turbo 10 — Turbo10 plan provided approx. 1000 kcal/d for all subjects and included portion controlled foods/shakes for the first week (week 0). All food, except non-starchy vegetables and no-calorie beverages, was provided for the first week (week 0). Starting week 1, subjects followed the My Way plan intervention through week 16.
  Arms: Nutrisystem Turbo 10
Behavioral: Nutrisystem My Way — The Nutrisystem My Way plan provided 7 breakfasts, 6 lunches, 6 dinners, and 7 (women) or 14 (men) snacks/desserts as pre-packaged portion controlled foods every week. Subjects were instructed to prepare one lunch and one dinner on their own each week. General guidelines and recommendations were provided by Nutrisystem in order to allow subjects to self-select appropriate foods for these eating occasions that fit within the My Way plan guidelines (~50% kcal from carbohydrate, ~25% from protein, ~25% from fat). Women were assigned to 1200 calories per day and men were assigned to 1500 calories per day. Nutrisystem packaged foods accounted for approximately 60% of daily calorie target; recommended grocery food additions (which subjects purchased on their own) accounted for the balance.
  Arms: Nutrisystem My Way
Behavioral: Nutrisystem DASH — The Nutrisystem DASH plan was a modification of the My Way plan designed to meet the nutrition profile of the DASH Diet, as described in NIH materials. Key nutritional targets included < 30% fat (< 7% saturated fat), < 150 mg/d of cholesterol, and < 2300 mg/d of sodium. Key dietary targets were consumption of 7-10 servings of fruit/vegetables/day, 2-3 servings of low-fat dairy/day, and 3 servings nuts/seeds/week. The Nutrisystem DASH plan included a subset of the Nutrisystem menu [7 breakfasts, 6 lunches, 6 dinners, plus snacks as portion-controlled foods every week], as well as modified guidelines for grocery additions, to achieve the nutrition targets of the DASH diet. Women consumed 1200 kcal/day and men consumed 1500 kcal/day.
  Arms: Nutrisystem DASH
Behavioral: Dieting on Your Own (DIY) - DASH — The self-directed diet included publicly available information consistent with the Dietary Approaches to Stop Hypertension (DASH) diet instructing individuals to consume a reduced calorie diet to support self-directed weight loss efforts. Women were assigned to a 1200 calorie diet and men were assigned to a 1500 calorie diet. Information on the self-directed diet was provided at the beginning of the intervention (visit 2, week 0). Subjects randomized to this group did not receive additional dietary counseling throughout the study period.
  Other Names: Self-directed Diet
  Arms: Dieting on Your Own (DIY) - DASH

SUMMARY:
The objective of this study was to determine changes in body weight and related outcomes achievable over a 16-week period in response to three different commercially available weight loss programs (Nutrisystem) providing pre-packed, portion controlled foods and beverages, each compared to a self-directed diet, in apparently healthy overweight and obese men and women.

DETAILED DESCRIPTION:
A randomized, controlled, four-arm parallel study design included two screening/baseline visits (visits 1 and 2; weeks -1 and 0) and six clinic visits (visits 3, 4, 5, 6, 7, 8, and 9; weeks 1, 2, 3, 4, 8, 12, and 16). One hundred and eighty healthy overweight and obese men and women (18-70 years of age; Body Mass Index 25.00 to 44.99 kg/m2) were randomly assigned (stratified randomization by two BMI and three age categories) to one of four treatment arms: a self-directed diet, or one of three different Nutrisystem programs: 1) My Way; 2) Turbo 10; or 3) a program modeled after the Dietary Approaches to Stopping Hypertension (DASH) diet. Daily energy intake targets for each 16-week intervention were 1500 kcal/day (men) or 1200 kcal/day (women), except for the first week of the Turbo 10 intervention, which included a more aggressive 1000 kcal/day diet to start. Body weight, body circumference (chest, waist, hip, upper arm, thigh and sum of the 5), and blood pressure measurements were obtained at baseline (week 0) and at weeks 1, 2, 3, 4, 8, 12, and 16 in the morning following an overnight fast (9 to 14 hours). Total and regional fat mass and fat-free mass (lean soft tissue and bone) were quantified by dual energy x-ray absorptiometry at baseline (week 0) and at weeks 4, 8, and 16. Analyses of serum lipoprotein lipids were obtained at baseline (week 0), week 8, and week 16. Lipoprotein lipid assessments included Total Cholesterol (TC), LDL-Cholesterol, HDL-Cholesterol, non-HDL-Cholesterol (calculated as TC minus HDL-C), Triglycerides, and the Total Cholesterol/HDL-Cholesterol ratio. Plasma chemistry and whole-blood hematology analyses were conducted at screening (week -1). Questionnaires designed to assess aspects of quality of life and sleep quality were administered at baseline (week 0) and weeks 4, 8, and 16. Quality of Life assessments included the Impact of Weight on Quality of Life-Lite (IQWOL-Lite), 36-Item Short Form Health Survey (SF-36), and Leeds Sleep Evaluation Questionnaire (LSEQ).

ELIGIBILITY:
Inclusion Criteria:

1. Subject is male or female, 18-70 years of age, inclusive.
2. Subject has a body mass index (BMI) of 25.00 to 44.99 kg/m2, inclusive, at visits 1 and 2 (weeks -1 and 0).
3. Subject has no plans to change smoking habits during the study period.
4. Subject is willing to follow study program instructions, including avoidance of all non-study-related food and beverages.
5. Subject is willing and able to comply with the visit schedule [i.e., no visit window will be allowed between visits 2 and 3 (week 0 and 1) and visits 3 and 4 (weeks 1 and 2)].
6. Subject agrees to follow the physical activity recommendations as outlined in each plan.
7. If a premenopausal female, subject has a history of regular menstrual cycles that range in length from 21 to 35 d, where applicable.
8. Judged to be in good health on the basis of medical history and screening laboratory assessments.
9. Subject understands the study procedures and signs forms providing informed consent to participate in the study and authorization for release of relevant protected health information to the study Investigators.

Exclusion Criteria:

1. Subject has an abnormal laboratory test result of clinical significance at visit 1 (week -1), at the discretion of the Investigator. One re-test will be allowed on a separate day prior to visit 2 (week 0) for subjects with abnormal laboratory test results.
2. Subject has had a weight loss or gain ≥10 lb (4.5 kg) in the 6 months prior to visit 1 (week -1).
3. Subject has used weight loss medications within 6 months of visit 1 (week -1) or weight loss supplements or programs, other than those provided, intended to alter body weight within 4 weeks of visit 1 (week -1) or during the course of the study (Appendix 1).
4. Subject has extreme dietary habits (e.g., Atkins diet, very high protein, vegetarian), in the opinion of the Investigator.
5. Subject has a known allergy, sensitivity, or intolerance to the study foods or any ingredients of the study menu provided.
6. Subject has diagnosed diabetes mellitus (type 1 or type 2) or fasting glucose ≥126 mg/dL at the screening visit (visit 1, week -1).
7. Subject has used thyroid hormones, except stable-dose replacement therapy for ≥2 months prior to visit 1 (week -1; Appendix 1).
8. Subject has used dietary supplements that, in the judgment of the Investigator, are likely to markedly affect appetite. The washout period will be 2 weeks prior to visit 1 (week -1; Appendix 1).
9. Subject has used medications or supplements that may influence carbohydrate metabolism, including but not limited to hypoglycemic medications and systemic (intravenous, intramuscular, or oral) or ≥1500 µg/d topical (inhaled, intranasal, or dermal) corticosteroids within 4 weeks of visit 1 (week -1) and throughout the study (Appendix 1).
10. Subject has a history or presence of clinically important cardiac, renal, hepatic, endocrine, pulmonary, biliary, pancreatic, or neurologic disorders.
11. Subject has an active gastrointestinal disorder such as peptic ulcer disease or malabsorption syndrome (mild lactose intolerance or gastroesophageal reflux diseases are acceptable).
12. Subject has an active infection or signs/symptoms of an infection. The baseline visit (visit 2, week 0) will be re-scheduled to allow subject to be symptom-free of any type of systemic infection for at least 5 days.
13. Subject has a history of gastrointestinal surgery for weight reducing purposes.
14. Subject has uncontrolled hypertension (systolic blood pressure ≥160 mm Hg or diastolic blood pressure ≥100 mm Hg as defined by the blood pressure measured at visit 1 (week -1). One re-test will be allowed on a separate day prior to visit 2 (week 0) for subjects whose blood pressure exceeds either of these cut points at visit 1.
15. Subject has a history or presence of cancer in the prior 2 years, except for non-melanoma skin cancer.
16. Subject is a female who is pregnant, planning to be pregnant during the study period, lactating, or is of childbearing potential and is unwilling to commit to the use of a medically approved form of contraception throughout the study period. The method of contraception must be recorded in the source document.
17. Subject is a premenopausal female using a form of hormonal contraception that does not result in a normal menstrual cycle, including a regular menses period.
18. Subject has a recent history of (within 12 months of visit 1, week -1) or strong potential for alcohol or substance abuse. Alcohol abuse defined as >14 drinks per week (1 drink = 12 oz beer, 5 oz wine, or 1½ oz distilled spirits).
19. Exposure to any non-registered drug product within 30 d prior to the screening visit (visit 1).
20. Individual has a condition the Investigator believes would interfere with his or her ability to provide informed consent, comply with the study protocol, or which might confound the interpretation of the study results or put the person at undue risk.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2015-04; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Body Weight | Up to 16 weeks
  Change in body weight from baseline (week 0) to each post-randomization visit (week 1, 2, 3, 4, 8, 12, and 16).

SECONDARY OUTCOMES:
Waist Circumference | Up to 16 weeks
  Change in waist circumference from baseline (week 0) to each post-randomization visit (week 1, 2, 3, 4, 8, 12, and 16).
Hip Circumference | Up to 16 weeks
  Change in hip circumference from baseline (week 0) to each post-randomization visit (week 1, 2, 3, 4, 8, 12, and 16).
Chest circumference | Up to 16 weeks
  Change in hip circumference from baseline (week 0) to each post-randomization visit (week 1, 2, 3, 4, 8, 12, and 16).
Upper arm circumference | Up to 16 weeks
  Change in upper arm circumference from baseline (week 0) to each post-randomization visit (week 1, 2, 3, 4, 8, 12, and 16).
Thigh circumference | Up to 16 weeks
  Change in thigh circumference from baseline (week 0) to each post-randomization visit (week 1, 2, 3, 4, 8, 12, and 16).
Body Weight (>=5%) | Up to 16 weeks
  percentage of subjects achieving at least a 5% loss of initial body weight from baseline (week 0) to each post-randomization visit (week 1,2,3,4,8,12, and 16)
Blood Pressure | Up to 16 weeks
  Change in systolic and diastolic blood pressure from baseline (week 0) to each post-randomization visit (week 1,2,3,4,8,12,16)
Quality of Life | Up to 16 weeks
  Change in IWQOL-Lite questionnaire subscale scores and total scores from baseline (week 0) to post-randomization visits 6,7, and 9 (week 4, 8, and 16).
Health Quality of Life | Up to 16 weeks
  Change in SF-36 questionnaire domain scores and composite score from baseline (week 0) to post-randomization visits 6,7, and 9 (week 4, 8, and 16).
Sleep Quality (questionnaire score) | Up to 16 weeks
  Change in sleep quality questionnaire score from baseline (week 0) to post-randomization visits 6,7, and 9 (week 4, 8, and 16).
Body Composition (Change in total fat mass) | Up to 16 weeks
  Change in total fat mass from baseline (week 0) to post-randomization visits 6,7, and 9 (week 4, 8, and 16).
Body Composition (Change in total fat free mass) | Up to 16 weeks
  Change in total fat free mass from baseline (week 0) to post-randomization visits 6,7, and 9 (week 4, 8, and 16).
Body Composition (Change in Android total fat mass) | Up to 16 weeks
  Change in Android total fat mass from baseline (week 0) to post-randomization visits 6,7, and 9 (week 4, 8, and 16).
Body Composition (Change in Gynoid total fat mass) | Up to 16 weeks
  Change in Gynoid total fat mass from baseline (week 0) to post-randomization visits 6,7, and 9 (week 4, 8, and 16).
Body Composition (Change in Abdominal Visceral total body fat) | Up to 16 weeks
  Change in Abdominal Visceral total body fat from baseline (week 0) to post-randomization visits 6,7, and 9 (week 4, 8, and 16).
Body Composition (Change in regional (trunk, non-trunk, arms and legs) total fat mass) | Up to 16 weeks
  Change in regional (trunk, non-trunk, arms and legs) total fat mass from baseline (week 0) to post-randomization visits 6,7, and 9 (week 4, 8, and 16).
Body Composition (Change in regional (trunk, non-trunk, arms and legs) total fat free mass) | Up to 16 weeks
  Change in regional (trunk, non-trunk, arms and legs) total fat free mass from baseline (week 0) to post-randomization visits 6,7, and 9 (week 4, 8, and 16).

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen M Kelley, MD, Principal Investigator — Biofortis Innovation Services; Chad M Cook, PhD, Study Director — Biofortis Innovation Services

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers.

REFERENCES:
- [Derived] Cook CM, McCormick CN, Knowles M, Kaden VN. A Commercially Available Portion-Controlled Diet Program Is More Effective for Weight Loss than a Self-Directed Diet: Results from a Randomized Clinical Trial. Front Nutr. 2017 Nov 7;4:55. doi: 10.3389/fnut.2017.00055. eCollection 2017. PMID 29164129